CLINICAL TRIAL: NCT02469324
Title: A Comparative RCT of Brief Internet-based Compassionate Mind Training and Cognitive-behavioral Therapy for Mothers and Their Babies
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: i4Health (Other)
Collaborators: Compassionate Mind Foundation (Unknown)
Responsible Party: Principal Investigator, Alex Kelman, PhD Candidate in Clinical Psychology - under the supervision of Alinne Barrera, PhD, Palo Alto University and i4Health, i4Health
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 15-018-H
Record Dates: First submitted 2015-06-05; First posted 2015-06-11 (Estimated); Last update posted 2016-02-23 (Estimated); Status verified 2016-02

CONDITIONS: Comparison of Internet-based CBT and CMT
MeSH Terms: interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cognitive-Behavioral Therapy (Active Comparator): see intervention explanation
  Interventions: Behavioral: Cognitive Behavioral Therapy
- Compassionate Mind Training (Experimental)
  Interventions: Behavioral: Compassionate Mind Training

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy — The course will be two weeks long, including the didactic portion of each course and the follow-up exercises (meditations for the CMT condition and exercises for the CBT condition) practiced daily for a total of two weeks. The course will contain two distinct parts. Part (a) will consist of a 45-minute didactic lesson that covers the basics of each approach. The course will provide a narrative rationale and the motivation for participants to complete the exercise portion of the course. Part (b) will be presented following completion of the didactic portion of the course. Participants will receive an automatically generated email following completion of the didactic that will include information on the follow-up exercises, suggestions for how to continue practicing, and a link to the the didactic portion of the course in case they want to review it again. Two weeks after enrollment and the completion of Part (b), participants will be invited to complete the post baseline measures.
  Arms: Cognitive-Behavioral Therapy
Behavioral: Compassionate Mind Training — see above
  Arms: Compassionate Mind Training

SUMMARY:
The current study is a two condition randomized controlled trial for women who are pregnant, interested in becoming pregnant, or pregnant within the last year. The conditions include a brief Cognitive Behavioral Therapy and a brief Compassionate Mind Training intervention. Participants in each condition will complete a 45 minute didactic exercises and readings followed by an email with exercises to continue practicing for a total of 2 weeks. After 2 weeks, participants will receive post-baseline assessment measures (e.g., depression, anxiety, affect, self-reassurance, self-attacking, self-criticizing, self-compassion). Participants will be recruited through a women's clinic in the United Kingdom by Michelle Cree, M.S. and through listservs by Yotam Heineberg, Psy.D. The researchers will also invite individuals in their social networks through email and through the Amazon Mechanical Turk System.

DETAILED DESCRIPTION:
The primary aim of this study is to provide support for the clinical utility of Internet-based Compassionate-Mind Training (CMT) with pregnant women, women who were recently pregnant, or women who are interested in becoming pregnant. Specifically, the investigators will compare an existing treatment, Internet-based Cognitive-Behavioral Therapy (CBT) psychoeducational resources to Internet-based CMT psychoeducational resources. The researchers hypothesize Internet-based CMT is more effective than Internet-based CBT in enhancing self-compassion and self-reassuring and decreasing self-criticizing and self-attacking. Additionally, the researchers hypothesize the CBT and CMT conditions will have near equivalence for improving participant affect as well as depression and anxiety.

An additional aim of the study is to assess the feasibility and acceptability of the course. As such, participants in each condition will be invited to complete the feedback questions for the course. The feedback questions will then be used in the hopes of adapting and improving the course based on participant feedback.

Up to 7.1% of new mothers in the United States may experience depression within the first three months of giving birth (Gavin et al., 2005). If minor depressive episodes are included, then the prevalence rate becomes as high as 19.2% (Gavin et al., 2005). The global incidence of postnatal depression is likely even higher (Almond, 2009). This course will target women who are interested in becoming pregnant, currently pregnant, or pregnant in the last year who seek to improve well-being during the perinatal period.

There is a strong base of research to suggest that maternal depression has significant impacts on offspring (Forman et al., 2007; Goodman, 2007). These effects tend to develop while the child is still in-utero (Forman et al., 2007; Goodman, 2007) and continue until the offspring reaches adulthood (Goodman & Brand, 2008). Research by Martins and Gaffan (2000) suggests that insecure attachment patterns are more common in children of depressed mothers than children of non-depressed mothers. Furthermore, insecure attachment style has substantial implications for persistent issues in functioning not only during childhood but throughout the entire lifespan (Martins & Gaffan, 2000). Since attachment is perhaps the most vital relationship during a human life, it is crucial to help make this relationship a positive one.

Of the PPD interventions analyzed in a meta-analysis by Clatworthy (2012), the briefest intervention was shown to positively impact PPD (Matthey, Kavanagh, Howie, Barnett, & Charles, 2004), whereas the longest intervention analyzed did not show an effect (Buist, Westley, & Hill, 1999). There is evidence to suggest that interventions based on psychological models are more effective than purely educational material (Clatworthy, 2012). Internet interventions, including the present course, have the advantages of being low cost while reaching large audiences around the world.

Nonconsumable interventions, or reusable interventions, are predominately automated and can be reused with minimal cost for each additional individual participant (Muñoz, 2010). Nonconsumable interventions are important for reducing health disparities worldwide, as they can be reused at low cost. The current Internet Intervention, which will aim to increase compassion, is both non-consumable and firmly grounded in the principles of Dr. Paul Gilbert's CFT. Additionally, the CFT condition will be compared to a CBT Internet intervention to assess relative efficacy. The researchers will focus specifically on the constructs of self-compassion, self-reassurance, self-attacking, depression, anxiety, and mood.

Self-compassion involves an individual being both aware and open to the internal suffering that one experiences (Neff, Hsieh, & Dejitterat, 2005), while keeping in mind that being imperfect is a trait shared across all humans (Neff & Vonk, 2009; Neff, 2009). Samaie and Farahani (2011) found that self-compassion served as a significant moderator between rumination and stress, suggesting that higher levels of self-compassion can decrease the relationship between rumination and stress (Samaie & Farahani, 2011). Also, self-compassion has also been linked to one's ability to balance one's own needs and the needs of another in a conflict situation (Yarnell & Neff, 2013). The cultivation of self-compassion has been shown to improve quality of shared decision making in interpersonal relationships as well as improve an individual's ability to balance her needs in a relationship with the needs of her partner (Yarnell & Neff, 2013).

CFT, which has an aim to increase compassion, is a movement towards a more biopsychosocial science of psychotherapy (Gilbert, 2010; Lawrence & Lee, 2013). It seeks to increase systemic harmony and ability to cultivate compassion for others, receive compassion from others, and direct compassion towards the self. This approach draws from social, developmental, evolutionary and Buddhist psychology (Gilbert, 2009). CFT holds that psychopathology manifests from unbalanced systems of affect regulation, such that the threat-based system is activated disproportionately to the contentment, safety, and soothing system. As such, this approach seeks to educate the participant about these systems and to increase the contentment, safety, and soothing system activity in order to augment compassion and well-being (Lawrence & Lee, 2013). Compassionate Mind Training (CMT) is the intervention component from the principles of CFT (Gilbert & Procter, 2006).

A lack of stimulation in the contentment, soothing, and safety system may also have physiological effects, particularly by inhibiting the production of oxytocin (Cree, 2010). When maternal oxytocin is disregulated, the parent-child bonding process can be adversely affected (Carter, 1998). Furthermore, irregularities in neuroendocrine activity related to attachment, history of the parent, and social atmosphere can make the bonding process more difficult (Carter, 2003). The use of CFT with a perinatal population has the ability to stimulate the aforementioned systems, improve the mother's compassion, and positively impact the attachment with her baby.

In a preliminary study, the researchers contacted participants from the UCSF Mothers and Babies Internet Project (Barrera, Kelman, & Muñoz, 2014). The majority of respondents stated they would be interested in learning how to be more compassionate (83% of English participants; 94% of Spanish participants). Also, these women asserted that Internet-based CMT would be useful to them (mean rating=7.41 out of 10).

The hypotheses of the current study are:

1. Following completion of the didactic portion of the course, participants will see greater increases in self-reassurance and decreases in self-attacking and self-criticizing in the CMT condition relative to the CBT condition.
2. Following completion of the didactic portion of the course, participants will see near equivalent affect improvements in the CMT and CBT conditions.
3. Following completion of the entire course, participants will see greater increases in self-compassion in the CMT condition relative to the CBT condition.
4. Following completion of the entire course, participants will see near equivalent reductions in depression and anxiety in the CMT and CBT conditions.

ELIGIBILITY:
Inclusion Criteria:

* Participants in the present study will include women over the age of 18 who are currently pregnant, pregnant within the last year, or endorse interest in becoming pregnant in the future. Additional inclusion criteria include proficiency in English and access to the Internet.

Exclusion Criteria:

* Exclusion criteria consist of not having interest in becoming pregnant, being male, or being under the age of 18.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2015-04; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
The Forms of Self-Criticizing/Attacking and Self-Reassurance Scale (FSCRS) | at baseline and following 45 minute didactic
  The Forms of Self-Criticizing/Attacking and Self-Reassurance Scale (FSCRS) will be administered to participants before and after the didactic portion of the course to assess change. This measure assesses levels of self-criticizing and attacking and capacity for self-reassurance (Gilbert, Clarke, Hempel, Miles, & Irons, 2004). The FSCRS is divided into three subscales: inadequate self, hated self, and reassured self. The items are on a Likert-Scale and there are five possible answers: "Not at all like me" (0 points); "A little bit like me" (1); "Moderately like me" (2); "Quite a bit like me" (3); and '"Extremely like me" (4). In a sample of female college students, Cronbach's alpha for inadequate self was at 0.90 and 0.86 for hated self and reassured self subscales (Gilbert et al., 2004).
Patient Health Questionnaire-4 (PHQ-4) | at baseline and following 2 week follow up
  The Patient Health Questionnaire-4 (PHQ-4) will be given to participants before the didactic portion of the course and following completion of the entire course to assess change. The PHQ-4 inventory consists of two self-report questions that measure depression through the PHQ-2 and two self-report questions that measure anxiety symptom severity through the GAD-2 (Kroenke, Spitzer, Williams, & Löwe, 2009). The items are on a Likert-Scale and there are four possible answers: "Not at all" (0 points); "Several days" (1); "More than half the days" (2); and "Nearly every day" (3). In the general population, Cronbach's alpha was .78 for PHQ-2 and .75 for GAD-2 (Löwe et al., 2010). When compared to SCID for DSM-IV diagnoses, a scaled score of 3 on the PHQ-2 scale demonstrated sensitivity of 87% and specificity of 78% for MDD, and it demonstrated comparable diagnostic performance relative to longer measures (Löwe, Kroenke, & Gräfe, 2005).
Self-Compassion Scale - Short Form (SCS-SF) | at baseline and following 2 week follow up
  The Self-Compassion Scale - Short Form (SCS-SF) will be given to participants before the didactic portion of the course and after completion of the entire course to assess change. Women who endorsed being "currently pregnant" at baseline will receive the SCS-SF again at 4-weeks postpartum to assess for any changes in self-compassion at this time. The SCS-SF measures how individuals respond to themselves during times of stress in order to assess level of self-compassion (Raes, Pommier, Neff, & Van Gucht, 2010). The items are on a Likert-Scale, and there are five possible answers that range from "Almost Never" (1 point) to "Almost Always (5)." The SCS-SF has a near perfect correlation with the longer version of the measure at .97. It has a Cronbach's alpha of .86 in the general population in the United States (Raes et al., 2010).
Participant Feedback Questionnaire (PFQ) | at 2 week follow up
  Participants from each condition will be invited to complete additional questionnaires regarding utilization of the course materials and the overall acceptability of the course to assess change. The Participant Feedback Questionnaires (PFQs) will include feedback on the number of times participants used the exercises and their overall impressions of the course materials.

CONTACTS AND LOCATIONS:
Overall Officials: Alex R Kelman, MS, Principal Investigator — Palo Alto University
Locations (1):
- Palo Alto University, Palo Alto, California, United States

REFERENCES:
- [Background] Gavin NI, Gaynes BN, Lohr KN, Meltzer-Brody S, Gartlehner G, Swinson T. Perinatal depression: a systematic review of prevalence and incidence. Obstet Gynecol. 2005 Nov;106(5 Pt 1):1071-83. doi: 10.1097/01.AOG.0000183597.31630.db. PMID 16260528
- [Background] Almond P. Postnatal depression: a global public health perspective. Perspect Public Health. 2009 Sep;129(5):221-7. doi: 10.1177/1757913909343882. PMID 19788165
- [Background] Forman DR, O'Hara MW, Stuart S, Gorman LL, Larsen KE, Coy KC. Effective treatment for postpartum depression is not sufficient to improve the developing mother-child relationship. Dev Psychopathol. 2007 Spring;19(2):585-602. doi: 10.1017/S0954579407070289. PMID 17459185
- [Background] Goodman SH. Depression in mothers. Annu Rev Clin Psychol. 2007;3:107-35. doi: 10.1146/annurev.clinpsy.3.022806.091401. PMID 17716050
- [Background] Goodman, S. H., & Brand, S. R. (2008). Parental psychopathology and its relation to child psychopathology. In Handbook of clinical psychology (pp. 937-965).
- [Background] Martins C, Gaffan EA. Effects of early maternal depression on patterns of infant-mother attachment: a meta-analytic investigation. J Child Psychol Psychiatry. 2000 Sep;41(6):737-46. PMID 11039686
- [Background] Clatworthy J. The effectiveness of antenatal interventions to prevent postnatal depression in high-risk women. J Affect Disord. 2012 Mar;137(1-3):25-34. doi: 10.1016/j.jad.2011.02.029. Epub 2011 Apr 22. PMID 21514960
- [Background] Matthey S, Kavanagh DJ, Howie P, Barnett B, Charles M. Prevention of postnatal distress or depression: an evaluation of an intervention at preparation for parenthood classes. J Affect Disord. 2004 Apr;79(1-3):113-26. doi: 10.1016/S0165-0327(02)00362-2. PMID 15023486
- [Background] Buist, A., Westley, D., & Hill, C. (1999). Antenatal prevention of postnatal depression. Archives of Women's Mental Health, 1(4), 167-173. doi:10.1007/s007370050024
- [Background] Munoz RF. Using evidence-based internet interventions to reduce health disparities worldwide. J Med Internet Res. 2010 Dec 17;12(5):e60. doi: 10.2196/jmir.1463. PMID 21169162
- [Background] Neff, K. D., Hsieh, Y.-P., & Dejitterat, K. (2005). Self-compassion, achievement goals, and coping with academic failure. Self and Identity, 4(3), 263-287. doi:10.1080/13576500444000317
- [Background] Yarnell, L. M., & Neff, K. D. (2013). Self-compassion, interpersonal conflict resolutions, and well-being. Self and Identity, 12(2), 146-159. doi:10.1080/15298868.2011.649545
- [Background] Neff KD, Vonk R. Self-compassion versus global self-esteem: two different ways of relating to oneself. J Pers. 2009 Feb;77(1):23-50. doi: 10.1111/j.1467-6494.2008.00537.x. Epub 2008 Nov 28. PMID 19076996
- [Background] Neff KD. The Role of Self-Compassion in Development: A Healthier Way to Relate to Oneself. Hum Dev. 2009 Jun;52(4):211-214. doi: 10.1159/000215071. No abstract available. PMID 22479080
- [Background] Samaie, G., & Farahani, H. a. (2011). Self-compassion as a moderator of the relationship between rumination, self-reflection and stress. Procedia - Social and Behavioral Sciences, 30, 978-982. doi:10.1016/j.sbspro.2011.10.190
- [Background] Lawrence VA, Lee D. An exploration of people's experiences of compassion-focused therapy for trauma, using interpretative phenomenological analysis. Clin Psychol Psychother. 2014 Nov-Dec;21(6):495-507. doi: 10.1002/cpp.1854. Epub 2013 Jul 24. PMID 23893917
- [Background] Gilbert, P. (2009). Introducing compassion-focused therapy. Advances in Psychiatric Treatment, 15(3), 199-208. doi:10.1192/apt.bp.107.005264
- [Background] Gilbert, P. (2010). The Compassionate Mind: A New Approach to Life's Challenges (p. 544). New Harbinger Publications.
- [Background] Gilbert, P., & Procter, S. (2006). Compassionate mind training for people with high shame and self-criticism: Overview and pilot study of a group therapy approach. Clinical Psychology and Psychotherapy, 13, 353-379. doi:10.1002/cpp
- [Background] Cree, M. (2010). Compassion focused therapy with perinatal and mother-infant distress. International Journal of Cognitive Therapy, 3(2), 159-171.
- [Background] Carter CS. Neuroendocrine perspectives on social attachment and love. Psychoneuroendocrinology. 1998 Nov;23(8):779-818. doi: 10.1016/s0306-4530(98)00055-9. PMID 9924738
- [Background] Barrera AZ, Kelman AR, Munoz RF. Keywords to recruit Spanish- and English-speaking participants: evidence from an online postpartum depression randomized controlled trial. J Med Internet Res. 2014 Jan 9;16(1):e6. doi: 10.2196/jmir.2999. PMID 24407163
- [Background] Carter CS. Developmental consequences of oxytocin. Physiol Behav. 2003 Aug;79(3):383-97. doi: 10.1016/s0031-9384(03)00151-3. PMID 12954433
- [Background] Lowe B, Kroenke K, Grafe K. Detecting and monitoring depression with a two-item questionnaire (PHQ-2). J Psychosom Res. 2005 Feb;58(2):163-71. doi: 10.1016/j.jpsychores.2004.09.006. PMID 15820844
- [Background] Lowe B, Wahl I, Rose M, Spitzer C, Glaesmer H, Wingenfeld K, Schneider A, Brahler E. A 4-item measure of depression and anxiety: validation and standardization of the Patient Health Questionnaire-4 (PHQ-4) in the general population. J Affect Disord. 2010 Apr;122(1-2):86-95. doi: 10.1016/j.jad.2009.06.019. Epub 2009 Jul 17. PMID 19616305
- [Background] Raes F, Pommier E, Neff KD, Van Gucht D. Construction and factorial validation of a short form of the Self-Compassion Scale. Clin Psychol Psychother. 2011 May-Jun;18(3):250-5. doi: 10.1002/cpp.702. Epub 2010 Jun 8. PMID 21584907
- [Derived] Kelman AR, Stanley ML, Barrera AZ, Cree M, Heineberg Y, Gilbert P. Comparing Brief Internet-Based Compassionate Mind Training and Cognitive Behavioral Therapy for Perinatal Women: Study Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2016 Apr 15;5(2):e65. doi: 10.2196/resprot.5332. PMID 27084301